CLINICAL TRIAL: NCT03839186
Title: The Effects of Anesthetic Drugs on Hemodynamic Changes in Cardiac Surgury and the Assotiation Between Gene Polymorphysim and Different Heart Diseases :a Pharmacogenetics Study
Brief Title: Pharmacogenetics Study on the Effects of Anesthetic Drugs on Circulatory Function
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XYHMZK PG 2000
Record Dates: First submitted 2017-12-13; First posted 2019-02-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2018-03

CONDITIONS: Drug Reaction; Anesthetic; Hemodynamic Rebound; Gene
Keywords: personalized medicine; genetic polymorphism; pharmacogenetics; hemodynamic change
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

SUMMARY:
This study intends to study the effects of anesthetics on Circulatory Function Genomics and find the anesthetic effects in pharmacodynamics, pharmacokinetics, drug receptor or target DNA level differences, further guiding individual treatment in clinic, promoting the development of precision the medicine.The anesthesia medication during perioperative period is more and more accurate,reasonable and safe, so as to improve the satisfaction of the patients and their families in the perioperative period, to ensure the safety of patients.

DETAILED DESCRIPTION:
This study is a non traumatic and non intervention study, and will use a large sample of clinical research, the number of subjects to be enrolled in the study group are 200 cases. The basic information of the study was included in the study before the operation. During the operation, the investigators need a collection of participants's arterial blood and monitor the hemodynamic index and anesthesia depth by bispectral index(BIS) . Further more，the investigators will follow up the participants' condition after operation.Dividing the patients into different groups according to their clinical features.The relationship between vital signs and the depth of anesthesia was analyzed and compared between different groups.Blood samples collected during the operation were detected by gene test. Comparing the results of genetic testing and clinical data analysis, then the investigators will find the differences in the expression of the gene polymorphisms of anesthetic drugs in the circulating function.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing general anesthesia
* Undergoing Cardiovascular surgery

Exclusion Criteria:

* ASA granding more than five
* Severe organ dysfunction

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from department of thoracic and cardiovascular surgery in Xiangya Hospital, Central South University
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Genotyping results of anesthetic drugs | one year
  Genotype information of SNP related to anesthetic drug metabolism, such as AA, AG or GG

SECONDARY OUTCOMES:
vital signs | one year
  The percentage of change in mean arterial pressure and heart rate

OTHER OUTCOMES:
depth of anesthesia | one year
  The value of BIS
prognostic indicator | one year
  The days of patients' hospital stay time

CONTACTS AND LOCATIONS:
Overall Officials: e wang, doctor, Study Chair — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No